CLINICAL TRIAL: NCT01595945
Title: Effect of Caloric Restriction and Gastric Bypass on Resting Metabolic Rate in Obese Subjects
Brief Title: Effect of Caloric Restriction and Gastric Bypass on Resting Metabolic Rate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: KiloCoach e.U. (Other)
Collaborators: Hospital Barmherzige Schwestern Vienna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KCKBHS-01
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
Keywords: Caloric restriction; Obesity; Gastric bypass; Resting metabolic rate
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gastric bypass (Other): Subjects with planned gastric bypass surgery are followed-up in regard of resting metabolic rate.
  Interventions: Procedure: Gastric bypass
- Caloric restriction (Other): Caloric restriction calculated by an online weight management program (based on subject's starting weight, start BMI, age, target weight and time span). Subjects are followed-up in regard to resting metabolic rate.
  Interventions: Behavioral: Caloric restriction

INTERVENTIONS:
Procedure: Gastric bypass — Subjects with a planned gastric bypass surgery are followed-up for resting metabolic rate.
  Arms: Gastric bypass
Behavioral: Caloric restriction — Subjects receive caloric restriction as calculated by an online weight management program and are followed-up for resting metabolic rate.
  Arms: Caloric restriction

SUMMARY:
Studies in overweight and obese subjects show a decline in resting metabolic rate (RMR) even after moderate caloric restriction. Yet the onset and course of such a metabolic adaption is still unclear. Lower resting metabolic rates were also reported after gastric banding bariatric surgery but have not yet been investigated in subjects after gastric bypass. The purpose of this study is to investigate the consequences on resting metabolic rate in subjects with obesity after moderate caloric restriction or gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30 kg/m2

Exclusion Criteria:

* Marked weight reduction in the last 2 years (>5% of initial body weight)
* Recent extreme fasting (during the last month)
* Manifest eating disorders (assignment to a specialist for eating disorders)
* Severe psychiatric disorders requiring treatment
* Pregnancy, lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Resting metabolic rate | 24 weeks

SECONDARY OUTCOMES:
Body composition (muscle mass, fat mass) | 24 weeks
Body Mass Index | 24 weeks
Caloric restriction | 24 weeks
Weight loss | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Aspalter, MD., Study Director — KiloCoach e.U.
Locations (2):
- Austria (2):
  - Hospital Barmherzige Schwestern Vienna, Vienna
  - KiloCoach e.U., Vienna